CLINICAL TRIAL: NCT02218190
Title: A Randomized Trial of Alvimopan for the Reduction of Ileus After Long Posterior Spinal Fusion
Brief Title: Alvimopan and Ileus in PSF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Orthopedic Research and Education Foundation (Other); Barnes-Jewish Hospital (Other)
Responsible Party: Principal Investigator, Michael Kelly, Assistant Prof. Department of Orthopedic Surgery, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201401126
Record Dates: First submitted 2014-08-13; First posted 2014-08-18 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Ileus; Spinal Fusion
Keywords: Alvimopan; Ileus; Posterior spinal fusion
MeSH Terms: conditions — Ileus | interventions — alvimopan; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alvimopan (Experimental): Alvimopan 12mg once orally two hours prior to surgery and then 2 mg orally twice a day until post-operative day (POD) seven.
  Interventions: Drug: Alvimopan
- Placebo - Sugar Pill (Placebo Comparator): Placebo Sugar Pill orally two hours prior to surgery and then one sugar pill orally twice a day until post-operative day (POD) seven
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alvimopan
  Other Names: Entereg
  Arms: Alvimopan
Drug: Placebo
  Other Names: Sugar Pill
  Arms: Placebo - Sugar Pill

SUMMARY:
The purpose of the study is to determine with Alvimopan reduces the incidence of post operative ileus in patients who undergo posterior spinal fusion.

DETAILED DESCRIPTION:
Posterior spinal fusion (PSF) is a common orthopaedic procedure associated with a high incidence of post-operative ileus (POI) and concomitant increased length of hospital stay (LOHS). POI is exacerbated by high dose opiate consumption often required by these patients post-operatively. We propose a randomized, double-blinded, placebo-controlled pilot trial studying the use of alvimopan, a peripherally-acting mu-opioid receptor antagonist known to reduce POI in bowel resection. We hypothesize that alvimopan will shorten POI in spine fusion patients without negatively affecting post-operative pain control. Treatment efficacy will be assessed by recording time to first bowel movement, time to hospital discharge, and post-operative pain control.

We hypothesize that acute administration of alvimopan, a peripherally-acting mu-opioid antagonist, shortens the duration of post-operative ileus (POI) in patients undergoing long-segment (5 or greater thoracolumbar levels) posterior spinal fusion (PSF). The study will be a randomized, double-blinded, placebo-controlled pilot trial. Reducing the morbidity of POI in patients undergoing PSF will decrease hospital stay and costs, and also improve patient satisfaction and post-operative care after major orthopaedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing elective PSF of at least 5 levels and/or fixation to pelvis

Exclusion Criteria:

* pregnant women
* ischemic heart disease
* chronic liver or renal disease
* prior bowel resection
* presence of colostomy or ileostomy
* gastroparesis
* complete bowel obstruction
* inflammatory bowel disease (ulcerative colitis or Crohn's disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Kelly, MD, Principal Investigator — Department of Orthopedic Surgery - Washington University in St. Louis School of Medicine
Locations (1):
- Barnes Jewish Hospital / Washington University in St. Louis School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Kehlet H, Holte K. Review of postoperative ileus. Am J Surg. 2001 Nov;182(5A Suppl):3S-10S. doi: 10.1016/s0002-9610(01)00781-4. PMID 11755891
- [Background] Senagore AJ. Pathogenesis and clinical and economic consequences of postoperative ileus. Am J Health Syst Pharm. 2007 Oct 15;64(20 Suppl 13):S3-7. doi: 10.2146/ajhp070428. PMID 17909274
- [Background] Leslie JB. Alvimopan for the management of postoperative ileus. Ann Pharmacother. 2005 Sep;39(9):1502-10. doi: 10.1345/aph.1E615. Epub 2005 Aug 2. PMID 16076918
- [Background] Holzer P. Opioids and opioid receptors in the enteric nervous system: from a problem in opioid analgesia to a possible new prokinetic therapy in humans. Neurosci Lett. 2004 May 6;361(1-3):192-5. doi: 10.1016/j.neulet.2003.12.004. PMID 15135926
- [Background] Kurz A, Sessler DI. Opioid-induced bowel dysfunction: pathophysiology and potential new therapies. Drugs. 2003;63(7):649-71. doi: 10.2165/00003495-200363070-00003. PMID 12656645
- [Background] Sternini C, Patierno S, Selmer IS, Kirchgessner A. The opioid system in the gastrointestinal tract. Neurogastroenterol Motil. 2004 Oct;16 Suppl 2:3-16. doi: 10.1111/j.1743-3150.2004.00553.x. PMID 15357847
- [Background] Behm B, Stollman N. Postoperative ileus: etiologies and interventions. Clin Gastroenterol Hepatol. 2003 Mar;1(2):71-80. doi: 10.1053/cgh.2003.50012. PMID 15017498
- [Background] Holte K, Kehlet H. Postoperative ileus: a preventable event. Br J Surg. 2000 Nov;87(11):1480-93. doi: 10.1046/j.1365-2168.2000.01595.x. PMID 11091234
- [Background] Zimmerman DM, Gidda JS, Cantrell BE, Schoepp DD, Johnson BG, Leander JD. Discovery of a potent, peripherally selective trans-3,4-dimethyl-4-(3-hydroxyphenyl)piperidine opioid antagonist for the treatment of gastrointestinal motility disorders. J Med Chem. 1994 Jul 22;37(15):2262-5. doi: 10.1021/jm00041a003. PMID 8057274
- [Background] Delaney CP, Weese JL, Hyman NH, Bauer J, Techner L, Gabriel K, Du W, Schmidt WK, Wallin BA; Alvimopan Postoperative Ileus Study Group. Phase III trial of alvimopan, a novel, peripherally acting, mu opioid antagonist, for postoperative ileus after major abdominal surgery. Dis Colon Rectum. 2005 Jun;48(6):1114-25; discussion 1125-6; author reply 1127-9. doi: 10.1007/s10350-005-0035-7. PMID 15906123
- [Background] Liu SS, Hodgson PS, Carpenter RL, Fricke JR Jr. ADL 8-2698, a trans-3,4-dimethyl-4-(3-hydroxyphenyl) piperidine, prevents gastrointestinal effects of intravenous morphine without affecting analgesia. Clin Pharmacol Ther. 2001 Jan;69(1):66-71. doi: 10.1067/mcp.2001.112680. PMID 11180040
- [Background] Viscusi ER, Goldstein S, Witkowski T, Andonakakis A, Jan R, Gabriel K, Du W, Techner L, Wallin B. Alvimopan, a peripherally acting mu-opioid receptor antagonist, compared with placebo in postoperative ileus after major abdominal surgery: results of a randomized, double-blind, controlled study. Surg Endosc. 2006 Jan;20(1):64-70. doi: 10.1007/s00464-005-0104-y. Epub 2005 Dec 7. PMID 16333556
- [Background] Wolff BG, Michelassi F, Gerkin TM, Techner L, Gabriel K, Du W, Wallin BA; Alvimopan Postoperative Ileus Study Group. Alvimopan, a novel, peripherally acting mu opioid antagonist: results of a multicenter, randomized, double-blind, placebo-controlled, phase III trial of major abdominal surgery and postoperative ileus. Ann Surg. 2004 Oct;240(4):728-34; discussion 734-5. doi: 10.1097/01.sla.0000141158.27977.66. PMID 15383800
- [Background] Buchler MW, Seiler CM, Monson JR, Flamant Y, Thompson-Fawcett MW, Byrne MM, Mortensen ER, Altman JF, Williamson R. Clinical trial: alvimopan for the management of post-operative ileus after abdominal surgery: results of an international randomized, double-blind, multicentre, placebo-controlled clinical study. Aliment Pharmacol Ther. 2008 Aug 1;28(3):312-25. doi: 10.1111/j.1365-2036.2008.03696.x. PMID 19086236
- [Background] Wolff BG, Viscusi ER, Delaney CP, Du W, Techner L. Patterns of gastrointestinal recovery after bowel resection and total abdominal hysterectomy: pooled results from the placebo arms of alvimopan phase III North American clinical trials. J Am Coll Surg. 2007 Jul;205(1):43-51. doi: 10.1016/j.jamcollsurg.2007.02.026. Epub 2007 May 17. PMID 17617331
- See also: Summary Review for Regulatory Action — https://www.accessdata.fda.gov/drugsatfda_docs/summary_review/2008/021775s000_sumr.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 Patients enrolled and withdrew prior to undergoing randomization, surgery and treatment
Groups:
- Alvimopan: Alvimopan 12mg once orally two hours prior to surgery and then 2 mg orally twice a day until post-operative day (POD) seven.
  Alvimopan
- Placebo - Sugar Pill: Placebo Sugar Pill orally two hours prior to surgery and then one sugar pill orally twice a day until post-operative day (POD) seven
  Placebo
Period: Overall Study
Arm/Group | Alvimopan | Placebo - Sugar Pill
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alvimopan | Placebo - Sugar Pill | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (17.5) | 54.7 (13.7) | 52.0 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 4 | 5 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Recovery of Bowel Function
Description: To determine the effect of alvimopan on the recovery of bowel function as determined by time to first bowel movement in patients undergoing posterior spinal fusion. The effect size calculated may guide a larger, multicenter randomized controlled study. Time was measured from wound closure to bowel movement.
Time Frame: 14 days or until hospital discharge whichever occurs first
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Alvimopan | Placebo - Sugar Pill
Number analyzed (Participants) | 13 | 13
Hours | 43.2 (23.1) | 34.0 (16.7)

2. Primary Outcome: Length of Hospital Stay
Description: To determine the effect of alvimopan on overall length of hospital stay in patients undergoing PSF.
Time Frame: 14 days or until hospital discharge whichever occurs first
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Alvimopan | Placebo - Sugar Pill
Number analyzed (Participants) | 13 | 13
Hours | 122.5 (48.4) | 117.2 (30.2)

3. Secondary Outcome: Complications and Adverse Event
Description: Number of patients with complication/adverse event.
Time Frame: 14 days or until hospital discharge, which ever occurs first
Measure: Count of Participants; unit: Participants
Arm/Group | Alvimopan | Placebo - Sugar Pill
Number analyzed (Participants) | 13 | 13
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 6 weeks after surgery.
Arm/Group | Alvimopan | Placebo - Sugar Pill
Serious Adverse Events (participants affected / at risk) | 2/13 | 3/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alvimopan (N=13) | Placebo - Sugar Pill (N=13)
Venothromboembolic Event (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Unrelated to intervention
Postoperative Hematoma (Surgical and medical procedures) | 1 (1) | 1 (1)
Screw malposition (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No